CLINICAL TRIAL: NCT04672434
Title: A Phase 1, Open-Label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Antineoplastic Activity of Sym024 (Anti-CD73) as Monotherapy and in Combination With Sym021 (Anti-PD-1) in Patients With Advanced Solid Tumor Malignancies
Brief Title: Sym024 Monotherapy and in Combination With Sym021 in Patients With Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Sym024-01
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Cancer; Solid Tumor
Keywords: Locally advanced/unresectable; Metastatic solid tumor; Anti-PD-1; PD-1; PD1; CD73; Squamous cell carcinoma of the head and neck (SCCHN); Non-small-cell lung carcinoma-adenocarcinoma histology subtype (NSCLC-Adeno); Pancreatic ductal adenocarcinoma (PDAC); Cholangiocarcinoma (CCA); Colorectal carcinoma (CRC); Gastric carcinoma (GC); Esophageal carcinoma (EsoCA); Mesothelioma (Meso); Sym021; Sym024; Head and neck squamous cell carcinoma (HNSCC); Cervical carcinoma (CC)
MeSH Terms: conditions — Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Cholangiocarcinoma; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Mesothelioma; Uterine Cervical Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Sym024 Dose Level 1 (Experimental): Part I, Sym024 monotherapy dose level 1
  Interventions: Drug: Sym024
- Sym024 Dose Level 2 (Experimental): Part I, Sym024 monotherapy dose level 2
  Interventions: Drug: Sym024
- Sym024 Dose Level 3 (Experimental): Part I, Sym024 monotherapy dose level 3
  Interventions: Drug: Sym024
- Sym024 Dose Level 4 (Experimental): Part I, Sym024 monotherapy dose level 4
  Interventions: Drug: Sym024
- Sym024 Dose Level -1 (Experimental): Part I, Sym024 monotherapy dose level -1. Evaluate only if needed based on tolerability
  Interventions: Drug: Sym024
- Sym021+Sym024 Dose Level 2 (Experimental): Part II, Sym021 in combination with dose level 2 of Sym024
  Interventions: Drug: Sym021; Drug: Sym024
- Sym021+Sym024 Dose Level 3 (Experimental): Part II, Sym021 in combination with dose level 3 of Sym024
  Interventions: Drug: Sym021; Drug: Sym024
- Sym021+Sym024 Dose Level 4 (Experimental): Part II, Sym021 in combination with dose level 4 of Sym024
  Interventions: Drug: Sym021; Drug: Sym024
- Sym021+Sym024 Dose Level 5 (Experimental): Part IIa, Sym024 monotherapy and in combination with Sym021
  Interventions: Drug: Sym021; Drug: Sym024
- Sym021+Sym024 Dose Level 1 (Experimental): Part II, Sym021 in combination with dose level 1 of Sym024. Evaluate only if needed based on tolerability
  Interventions: Drug: Sym021; Drug: Sym024
- Dose Expansion Sym021 (+Sym024) (Experimental): Part III, dose expansion Sym024 and/or Sym021+Sym024
  Interventions: Drug: Sym021; Drug: Sym024

INTERVENTIONS:
Drug: Sym021 — Sym021 is a humanized anti-PD-1 antibody.
  Other Names: Anti-PD-1
  Arms: Dose Expansion Sym021 (+Sym024); Sym021+Sym024 Dose Level 1; Sym021+Sym024 Dose Level 2; Sym021+Sym024 Dose Level 3; Sym021+Sym024 Dose Level 4; Sym021+Sym024 Dose Level 5
Drug: Sym024 — Sym024 is an anti-CD73 antibody.

SUMMARY:
The primary purpose of this study is to see if Sym024 is safe and tolerable as monotherapy and in combination with Sym021 in patients with solid tumor malignancies.

DETAILED DESCRIPTION:
Part 1 of this study will assess the safety and tolerability to establish the maximum tolerated dose (MTD) (or the maximum administered dose [MAD]) and/or the selected dose(s) of Sym024 in patients with solid tumor malignancies.

Part 2 of this study will assess the safety and tolerability to establish the MTD (or the MAD) and/or the selected dose(s) of Sym024 when administered in combination with Sym021 in patients with solid tumor malignancies.

Part 2a of this study will assess the safety and tolerability of Sym024 when first administered as a single agent during Cycle 1 (safety lead-in) followed by administration in combination with Sym021 during Cycle 2 and subsequent cycles.

Part 3 of this study will assess the safety of Sym024 when administered alone or in combination with Sym021 in expanded cohorts of patients with solid tumor malignancies.

April 2024: The above was the study design at trial start. Per protocol, implementation of a part 3 would require an amendment. However, this was never done as it was decided not to include a part 3.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥18 years.
* Documented (histologically or cytologically proven), locally advanced or metastatic solid tumor malignancy (must be one of the following):

  1. Squamous cell carcinoma of the head and neck
  2. Non-small-cell lung carcinoma-adenocarcinoma histology subtype
  3. Pancreatic ductal adenocarcinoma
  4. Cholangiocarcinoma
  5. Colorectal carcinoma (microsatellite stable [MSS] and microsatellite instability-high [MSI-H] phenotypes)
  6. Gastric carcinoma (includes gastroesophageal carcinoma)
  7. Esophageal carcinoma (includes squamous cell and adenocarcinoma)
  8. Mesothelioma (pleural and peritoneal)
  9. Cervical carcinoma (CC) (includes adeno, squamous and mixed adeno-squamous carcinoma histology subtypes)
* Malignancy that is not currently amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
* Measurable disease according to RECIST v1.1.
* Refractory to or intolerant of existing therapy(ies) known to provide clinical benefit.
* Agreeing to mandatory tumor tissue biopsies (2 total).
* ECOG PS of 0 or 1.
* Adequate organ function as indicated by the following laboratory values.
* Adequate contraception required as appropriate.

Exclusion Criteria:

* Central nervous system (CNS) malignancies.
* Clinically significant cardiovascular disease or condition.
* Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism within 4 weeks prior to the first dose of study drug(s).
* Active uncontrolled bleeding or a known bleeding diathesis.
* Significant ocular disease or condition.
* Significant pulmonary disease or condition.
* Current or recent (within 6 months) significant gastrointestinal disease or condition.
* Active, known or suspected autoimmune disease.
* History of organ transplantation (i.e., stem cell or solid organ transplant).
* Known history of human immunodeficiency virus (HIV) or known active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Any other serious/active/uncontrolled infection.
* History of significant toxicities associated with previous administration of immune checkpoint inhibitors.
* Known or suspected hypersensitivity to any of the excipients of formulated study drug.
* Unresolved >Grade 1 toxicity associated with any prior antineoplastic therapy.
* Inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to the first dose of study drug(s).
* Any other serious, life-threatening, or unstable preexisting medical condition (aside from the underlying malignancy).

Therapeutic Exclusions

* Prior therapy with Sym024 or other inhibitors of CD73, CD39 or adenosine receptors ADORA2A, ADORA2B.
* Part II and Part III, prior anti-PD-(L)1 therapy, except for indications where it is approved.
* Any antineoplastic agent for the primary malignancy (standard or investigational) within 4 weeks or 5 elimination half-lives.
* Any other investigational treatments within 2 weeks prior to the first dose of study drug(s).
* Radiotherapy, with exceptions.
* Live vaccines against infectious diseases 4 weeks prior to the first dose of study drug(s).
* Immunosuppressive or systemic glucocorticoids therapy (>10 mg daily prednisone or equivalent) within 2 weeks prior to the first dose of study drug(s), with exceptions.
* Prophylactic use of hematopoietic growth factors within 1 week prior to the first dose of study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Part I: To evaluate the incidence, severity and relationship of (S)AEs to establish the MTD/MAD of Sym024 monotherapy. | 28 days
  Assess the safety and tolerability of Sym024 monotherapy on a Q2W schedule (every two weeks). Assessment based on the occurrence of AEs meeting DLT criteria measured during Cycle 1
Part II: To evaluate the incidence, severity and relationship of (S)AEs to establish MTD/MAD of Sym024 in combination with Sym021. | 28 days
  Assess the safety and tolerability of the sequential escalating doses of Sym024 in combination with Sym021 on a Q2W schedule. Assessment based on the occurrence of AEs meeting DLT criteria measured during Cycle 1
Part III: To evaluate the incidence, severity and relationship of (S)AEs to further assess safety of Sym024 when administered alone or in combination with Sym021. | 12 months
  Assess the safety and tolerability of Sym024 and/or Sym021+Sym024 on a Q2W schedule. Assessment based on the occurrence of AEs

SECONDARY OUTCOMES:
Evaluation of the immunogenicity of Sym024 as a single agent and in combination with Sym024 | 24 months
  Serum sampling to assess the potential for anti-drug antibody (ADA) formation
Evaluation of objective response (OR) or stable disease (SD) | 24 months
  Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST)
Time to progression (TTP) of disease | 24 months
  Based on time of enrollment to first evidence of progression on imaging studies, as assessed by RECIST v1.1 and iRECIST
Area under the concentration-time curve in a dosing interval (AUC) | 24 months
  Will be estimated using non-compartmental methods and actual timepoints
Maximum concentration (Cmax) | 24 months
  Will be derived from observed data
Time to reach maximum concentration (Tmax) | 24 months
  Will be derived from observed data
Trough concentration (Ctrough) | 24 months
  Will be derived from observed data
Terminal elimination half-life (T½) | 24 months
  Will be estimated using non-compartmental methods and actual timepoints
Clearance (CL) | 24 months
  Will be estimated using non-compartmental methods and actual timepoints

CONTACTS AND LOCATIONS:
Overall Officials: N. Lakhani, MD PhD, Principal Investigator — START Midwest, USA
Locations (4):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No